CLINICAL TRIAL: NCT06127303
Title: A Single-arm, Phase II Clinical Study of Toripalimab Combined With Cryoablation for First-line Oligo-progression in Driver-negative Advanced NSCLC
Brief Title: Toripalimab Combined With Cryoablation for First-line Oligo-progression in Driver-negative Advanced NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Ziming Li, Deputy Director, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS23070
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Oligo-progression; Toripalimab; Cryoablation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab; Immunotherapy; Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Toripalimab Combined with Cryoablation (Experimental): Patients with oligometastatic driver-negative advanced NSCLC after first-line immunotherapy progress would be treated with Toripalimab Combined with Cryoablation.
  Interventions: Drug: Toripalimab; Other: Cryoablation

INTERVENTIONS:
Drug: Toripalimab — Toripalimab treatment (240mg intravenously every 3 weeks) started on day 3 after cryoablation, until occurrence of termination event specified in the protocol.
  Other Names: Immunotherapy
Other: Cryoablation — The ablation was performed on the first day of each cycle, and the target lesions were comprehensively screened for cryoablation based on the location and size of the lesions.

SUMMARY:
Immunotherapy with programmed death-1(PD-1) inhibitors is now standard therapy for first-line use in patients with driver-negative advanced NSCLC, whether as single-agent or in combination with chemotherapy. After progression of first-line immunotherapy, NSCLC patients may be treated with chemotherapy, radiotherapy or targeted therapies, among others. Recently, Immune Checkpoint inhibitors (ICIs) rechallenge has become a highly anticipated option. Although the objective response rate of the ICIs rechallenge patients has decreased substantially compared with the efficacy of the first ICI treatment, nearly 50% of patients can regain disease control.

Cryoablation is a minimally invasive technique that utilizes very low temperature to eliminate viable tumour cells in target tissues. It has been reported that ablation can enhance immune response.

The objective of this study was to evaluate the efficacy and safety of toripalimab (PD-1) in combination with cryoablation in the treatment of oligometastatic driver-negative advanced NSCLC after first-line immunotherapy progress.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation and written informed consent;
* histologically or cytologically confirmed advanced metastatic (stage IV) non-small cell lung cancer;
* Patients with negative driver genes who develop oligoprogression after receiving standard first-line therapy. The oligoprogression is defined as: 1-5 metastatic lesions, and no more than 3 organs;
* Age 18-75 years old; ECOG PS: 0-1; The expected survival is more than 3 months;
* At least one measurable lesion;
* Patients were willing to provide adequate blood and tissue samples；
* Patients had adequate hematologic, renal, and liver function;
* International normalised ratio (INR) ≤1.5 and partial thromboplastin time (PTT or aPTT) ≤1.5 x ULN within 7 days prior to study treatment;
* The woman patients of childbearing age who must agree to take contraceptive methods during the research;
* The man patients who must agree to take contraceptive methods during the research and within another 6 months after it.

Exclusion Criteria:

* cytologically or histologically confirmed combination with small cell lung cancer component or sarcomatoid element;
* Previously received targeted therapy for advanced NSCLC (including osimertinib, erlotinib, crizotinib, etc);
* Had undergone major surgical operations or had not fully recovered from previous operations within 3 weeks before enrollment;
* Known active nervous system (CNS) metastases and/or carcinomatous meningitis;
* Spinal cord compression for which operation and/or radical radiotherapy has not been given, or no clinical evidence of stable disease for ≥4 weeks prior to enrollment after treatment for previously diagnosed spinal cord compression;
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage; patients with stable symptoms after drainage can be enrolled;
* History of idiopathic pulmonary fibrosis, organized pneumonia (e.g., obliterating bronchiolitis), drug induced pneumonia, idiopathic pneumonia or evidence of active pneumonia during chest CT scanning for screening;
* Clinically uncontrolled active infection, including but not limited to acute pneumonia;
* Uncontrollable major epileptic seizure or superior vena cava syndrome;
* Previous or current co-occurrence of other malignancies (excluding controllable non-melanoma basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the breast or cervix, superficial bladder cancer, or other carcinoma in situ);
* Known hepatic diseases of clinical significance, including active viral hepatitis, alcoholic hepatitis or other hepatitis, liver cirrhosis, fatty liver, hereditary liver disease;
* Active tuberculosis (TB), receiving anti-tuberculosis therapy currently or within one year prior to screening;
* Use of systemic immunosuppressive therapy for any active autoimmune disease within two years prior to Day 1 of the 1st cycle;
* Vaccination of live-virus vaccine within 30 days after the start of planned treatment; Inactivated seasonal influenza vaccine was permitted;
* Patients has HIV-positive;
* Patients judged by the investigator to be inappropriate as a subject of this study.
* History of severe allergic, quasi-allergic, or other hypersensitive reactions to chimeric or humanized antibodies or fusion proteins;
* Known allergy to biological drugs produced from Chinese hamster ovary cells, or to citrate monohydrate, sodium citrate dihydrate, mannitol, polysorbate (components of the study drug);
* Patients who have previously received allogeneic stem cells or parenchymal organ transplants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2028-04-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 6 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or date of death, whichever occurred first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on RECIST 1.1.
Disease control rate (DCR) | 6 months
  DCR was defined as the percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable.
Overall Survival (OS) | 24 months
  OS was defined as the duration from the date of randomization until the date of death from any cause.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 2 years
  Frequency table will be used to summarize occurrence of each treatment-emergent AE. Number and classification of participants with treatment-related adverse events as assessed by CTCAE v5.0 were recorded.
Correlation analysis of PD-L1 expression of tumor and ORR | Up to 1 years
  Correlation Analysis of the PD-L1 expression in tumor tissue specimen related with the tumor response.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No